CLINICAL TRIAL: NCT00925392
Title: Doripenem Intrapulmonary Pharmacokinetics in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keith A. Rodvold (Other)
Collaborators: Pulmonary Associates, PA (Unknown)
Responsible Party: Sponsor-Investigator, Keith A. Rodvold, Professor, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DORICPK4002
Record Dates: First submitted 2009-06-17; First posted 2009-06-22 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: doripenem; epithelial lining fluid; alveolar macrophages; pharmacokinetics; Healthy adult subjects
MeSH Terms: interventions — Doripenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doripenem 500 mg (Experimental)
  Interventions: Drug: Doripenem
- Doripenem 1000 mg (Experimental)
  Interventions: Drug: Doripenem

INTERVENTIONS:
Drug: Doripenem — Intravenous 500 mg every (q) 8 hours for 3 doses
  Other Names: Doribax
  Arms: Doripenem 500 mg
Drug: Doripenem — Intravenous 1000 mg q 8 hours for 3 doses
  Other Names: Doribax
  Arms: Doripenem 1000 mg

SUMMARY:
This study is being performed to measure the amount of the antibiotic doripenem (study drug) found in the fluid and cells of the lung and blood after receiving three doses of doripenem. The major objectives of this research are to see how much and for how long doripenem gets into the fluids and cells of the lungs of healthy adult subjects.

DETAILED DESCRIPTION:
The primary objective of this descriptive study is to determine and compare the plasma, epithelial lining fluid (ELF), and alveolar macrophages (AM) concentrations following multiple intravenous doses of doripenem in healthy, non-smoking adult subjects. In brief, each subject who qualifies for the study will be randomized to one of two dosing regimens: doripenem 500 mg or doripenem 1000 mg every 8 hours for a total of three intravenous doses. Each dose of doripenem will be administered as an intravenous infusion over 4 hours. Serial blood samples for determining plasma doripenem concentrations will be collected prior to and after the start of the intravenous infusion of the third doripenem dose. Each subject will undergo one standardized bronchoscopy with BAL in the outpatient bronchoscopy suite at one of four sampling times after the start of the intravenous infusion of the third doripenem dose. BAL collection will provide samples to determine drug concentration in ELF and AM. Safety will be assessed throughout the study by adverse event monitoring, clinical laboratory tests, and vital sign monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women at least 18 years of age who have no history of smoking within the last 1 year.
* Subjects must be healthy with no clinically important abnormalities in the medical history, physical examination, or laboratory values.

Exclusion Criteria:

* Subjects must not have a history of allergic or other serious reactions to doripenem or any beta-lactam antibiotic, benzodiazepines or lidocaine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine and compare the plasma, epithelial lining fluid, and alveolar macrophages concentrations following multiple intravenous doses of doripenem in healthy, non-smoking adult subjects. | 32 hours

SECONDARY OUTCOMES:
The secondary objective of this study is the assessment of safety and tolerability of doripenem as measured by the overall incidence of treatment-emergent adverse events. | 24 hours post end of doripenem administration

CONTACTS AND LOCATIONS:
Overall Officials: Keith A. Rodvold, Pharm.D., Principal Investigator — University of Illinois at Chicago; Larry H. Danziger, Pharm.D., Principal Investigator — University of Illinois at Chicago; Mark H. Gotfried, M.D., Principal Investigator — Pulmonary Associates, PA
Locations (1):
- Pulmonary Associates, PA, Phoenix, Arizona, United States